CLINICAL TRIAL: NCT04322214
Title: Clinical Trial to Evaluate Pharmacological Interactions Between γ-hydroxybutyrate (GHB) and Cobicistat
Acronym: GHB_Cobi
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: GHB_Cobi; 2019-002122-71 (EudraCT Number)
Record Dates: First submitted 2019-12-10; First posted 2020-03-26 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Pharmacokinetic Interactions; HIV
Keywords: pharmacokinetic interactions; chemsex; GHB; cobicistat; γ-hydroxybutyrate
MeSH Terms: conditions — Chemsex | interventions — Cobicistat; Sodium Oxybate

STUDY DESIGN:
Intervention Model Description: Participants will undergo two 5-day treatment periods (COBI and placebo) separated by a 7-day washout period:
  * COBI period: volunteers will receive once daily cobicistat (150 mg QD) for 5 days.
  * Placebo period: volunteers will receive once-daily placebo (lactose) for 5 days. On day 5 of each treatment period, participants will receive a single oral dose of GHB (25 mg/kg).
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COBI period (5 days) + Placebo period (5 days) (Experimental): volunteers will receive once daily cobicistat for 5 days. On day 5, participants will receive a single oral dose of GHB. After a washout period for 7 days, volunteers will receive once-daily placebo for 5 days. On day 5, participants will receive a single oral dose of GHB
  Interventions: Drug: Cobicistat 150 MG; Drug: Placebo; Drug: GHB
- Placebo period (5 days) + COBI period (5 days) (Experimental): volunteers will receive once-daily placebo for 5 days. On day 5, participants will receive a single oral dose of GHB. After a washout period for 7 days, volunteers will receive once daily cobicistat for 5 days. On day 5, participants will receive a single oral dose of GHB.
  Interventions: Drug: Cobicistat 150 MG; Drug: Placebo; Drug: GHB

INTERVENTIONS:
Drug: Cobicistat 150 MG — once daily cobicistat (150 mg QD) for 5 days
  Other Names: Cobicistat
Drug: Placebo — once daily lactose capsules (as aspect cobicistat capsules)
Drug: GHB — single oral dose of GHB (25 mg/kg) on days 5 and 17
  Other Names: XYREM

SUMMARY:
Gamma-hydroxybutyric acid (GHB) is a popular "party drug" because it is inexpensive and easy to ingest. The calming and euphoric effects of GHB in low doses have given the drug the nickname "liquid ecstasy". However, at doses >60 mg/kg coma, convulsions, and respiratory depression can occur. If the drug combinates with alcohol these effects intensify, especially respiratory depression and hypotension.

Lately a phenomenon called Chemsex has been spreading across big European cities. This is a form of recreational drug use and it is believed that can be, in part, the cause of the increasing in consumption of GHB. Chemsex is especially common among men who have sex with other men (MSM) and in people living with HIV, with up to 50% of HIV-positive MSM reporting to be engaged in chemsex in recent months. This population is specially concerning since the combination of ART with the drug can cause pharmacological interactions leading to overdose.

Specifically, this study intends to evaluate the drug interaction with low doses of cobicistat, an antiretroviral drug enhancer, since there are two case reports of life-threatening overdoses in patients on treatment with high doses of another enhancer that has a similar effect than cobicistat, but there are no studies about interactions with low doses.

DETAILED DESCRIPTION:
Gamma-hydroxybutyric acid (GHB) is an endogenous compound present in most mammalian tissues at nanomolar concentrations and a minor metabolite or precursor of gammaaminobutyric acid (GABA). GHB was first synthesized in 1960 by the French biochemist H.-M. Laborit who was searching for analogues of GABA. Currently, medically formulated GHB sodium oxybate (Xyrem®) is approved in different countries for such varied uses as general anaesthesia, the treatment of alcohol withdrawal and addiction, and cataplexy associated with narcolepsy.

Pharmacokinetics of GHB are characterized by rapid oral absorption, with peak concentrations in plasma 20-45 min after dosing, and half-life of 20-30 min. The majority of the dose is eliminated completely within 4-8 h. Metabolism of GHB occurs via GHB dehydrogenase, which transforms it into succinic semialdehyde and, by a second oxidation step with transformation into succinic acid, it is then ultimately metabolized to water and excreted through breath as carbon dioxide. However, GHB exposure is increased in patients with liver function impairment and has been suggested presystemic (hepatic first pass) metabolism mediated by the CYP450 system in humans.

During the 1980s, easy access to GHB-containing products led to various unapproved uses, including weight loss, bodybuilding and the treatment of sleeplessness, sometimes with serious long-term effects. During the last years, GHB has become a major concern in emergency rooms of some countries due to an important increase in the number of cases of intoxications.

Since the drug is both inexpensive and easy to ingest, it has been popular as a "party drug." The calming and euphoric effects of GHB in low doses (20-30 mg/kg) have given the drug the nickname "liquid ecstasy". At higher doses (> 50 mg/kg), the hypnotic effects are more prominent and at doses >60 mg/kg coma, convulsions, and respiratory depression can occur. The clinical hallmark of GHB poisoning is rapid onset of coma, with respiratory depression, hypoventilation and bradycardia. Combination with alcohol potentiates these effects, especially respiratory depression and hypotension.

Regular use of GHB is thought to be relatively higher in the lesbian, gay, bisexual, and transgender community. Anecdotal evidence suggests that GHB use is increasing and this may be driven in part by an increase in the incidence of chemsex. Chemsex is a specific form of recreational drug use involving specific drugs such as GHB/γ-butyrolactone (GBL), methylamphetamine and mephedrone, alone or in combination, to enhance or prolong sexual sessions. Such sessions can last for several days, involve multiple partners and include high risk behaviour.

Although the phenomenon of chemsex was initially limited to the metropolitan area of London, it is getting spread across other big European cities, making of this an emerging global health issue. Chemsex is especially common among men who have sex with other men (MSM) and in people living with HIV (PLWH), with up to 50% of HIV-positive MSM reporting to be engaged in chemsex in recent months.

Consumption of recreational drugs in PLWH has been associated with high-risk practices for sexually transmitted diseases. In addition, use of drugs in patients taking antiretroviral therapy (ART) might result in pharmacological interactions with potential risk of overdosing. Noteworthy, widespread use of chemsex drugs has resulted in increased rates of overdose and associated deaths, and Handley & Flanagan have reported an increase in the number of cases of fatal poisoning with GHB, mephedrone and ketamine in England and Wales since 2008. Also, GHB-associated deaths have been reported from the USA, Canada, Europe and Australia.

Cobicistat (GS-9350) is a pharmacokinetic enhancer that was developed to inhibit CYP3A activity in a time- and concentration-dependent manner, thus boosting other antiretroviral drugs. Results from clinical trials showed that it can increase the plasma exposure of elvitegravir, atazanavir, and darunavir. Similarly, cobicistat increases the exposure to many other xenobiotics. For example, it is well known that CYP3A4 inhibition leads to a significant increase in concentrations of sildenafil and other erectile dysfunction agents, and that a dose adjustment is needed in this scenario. Similarly, CYP3A4 inhibition increased ketamine exposure in a small clinical trial in healthy volunteers.

There are two case reports in the literature of well documented life-threatening overdoses on GHB and MDMA in HIV-positive patients on treatment with high-doses of ritonavir (600 mg bid). However, the possibility for this drug interaction with the low doses of pharmacoenhancers currently used (ritonavir 100 mg qd, cobicistat 150 mg qd) is still a matter for debate, Despite data suggesting the possibility of drug interactions between cobicistat and GHB, formal pharmacokinetic studies assessing this issue are lacking.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females* aging 18-45 years.
2. Body weight ranging between 50 and 100 Kg.
3. Previous experience with the consumption of sedatives (alcohol, cannabis, benzodiazepines, GHB or other hypnotics).
4. Absence of abnormalities in the screening ECG and blood/urine tests.
5. Agree with the study procedures and signature of the informed consent.

   * Women of childbearing potential must have a negative pregnancy test prior to randomization into the study and commitment to use at least one of these birth control methods: male or female condom with or without spermicide, cap, diaphragm or sponge with or without spermicide, intrauterine device, bilateral tubal occlusion, vasectomized partner, sexual abstinence during the study. Condom use is considered as an additional method of contraception only and cannot be the only method of contraception used as not been considered an effective method by the Clinical Trial Facilitation Group (CTFG) guidelines.

Based on ICH, M3 (R2) 2009 a woman is considered of childbearing potential: fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include tubal ligation, hysterectomy, bilateral oophorectomy.

Exclusion Criteria:

1. Prior history of medical or psychiatric adverse reaction following GHB consumption.
2. Current substance use disorder (DSM-V, dependence, addiction) of any drug or substance of abuse.
3. Prior history of substance use disorder (DSM-V, drug use disorder or addiction) of any drug or substance of abuse (except nicotine).
4. Smokers>10 cigarettes/day.
5. History of any physical condition or major surgery within the previous three months.
6. History of individual psychiatric conditions or schizophrenia in first-degree relatives.
7. History of gastrointestinal, hepatic, renal diseases or other conditions which, in opinion of the investigator, may affect drug absorption, distribution, metabolism or elimination.
8. Alcohol intake higher than 4 units/day (40 g) in men or 2 units/day (20 g) in women.
9. Positive urine drug test (Amphetamines, Barbiturates, Benzodiazepines, Cocaine, MDMA, Methamphetamine, Morphine/Opioids, Methadone, tricyclic antidepressants, THC)
10. HIV infection, chronic hepatitis C (IgG VHC) or B (HBsAg).
11. Lactose intolerance
12. Pregnancy, lactation, or planned pregnancy during the study period.
13. Current or recent pharmacological treatment (≥3 doses per week) in the last 2 weeks
14. Blood donation in the 3 previous months
15. Participation in another clinical trial in the previous 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
concentration in plasma of GHB | days 5 and 17
  mg/dl
Proportion of participants reporting adverse events. | Since baseline to day 28
  % of participants developing related adverse events.

SECONDARY OUTCOMES:
physiological effects: blood pressure | days 5 and 17
  mmHg
physiological effects: heart rate | days 5 and 17
  lat/min
physiological effects : oxygen saturation | days 5 and 17
  percentage (%)
subjective effects of GHB -ARCI | days 5 and 17
  Addiction Research Center Inventory (ARCI) 49 item short for questionnaire (measures sedation, euphoria, dysphoria, energy and stimulation)
subjective effects of GHB - Visual analog scale | days 5 and 17
  visual analog scales (VAS) 15 items (about sensations (good or bad), feelings, nausea and vomit) determined by horizontal line of 100 mm. The ends are defined as the limits of the parameter to be measured orientated from the left (minimum intensity) to the right (maximum intensity).

CONTACTS AND LOCATIONS:
Overall Officials: José Moltó, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- José, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Molto J, Bailon L, Perez-Mana C, Papaseit E, Miranda C, Martin S, Mothe B, Farre M. Absence of drug-drug interactions between gamma-hydroxybutyric acid (GHB) and cobicistat. J Antimicrob Chemother. 2021 Dec 24;77(1):181-184. doi: 10.1093/jac/dkab359. PMID 34561695